CLINICAL TRIAL: NCT06777537
Title: Neoadjuvant Chemotherapy with or Without Talniflumate for the Treatment of Breast Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Qifeng Yang, Professor, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HECT005
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — talniflumate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Talniflumate (Experimental): Patients will be treated with adjuvant treatment . And Talniflumate will be administrated.
  Interventions: Drug: Talniflumate
- Placebo (No Intervention): Patients will be treated with Placebo

INTERVENTIONS:
Drug: Talniflumate — Talniflumate was administered
  Arms: Talniflumate

SUMMARY:
RATIONALE:

Talniflumate, a prodrug of niflumic acid with significant anti-inflammatory properties, has emerged as a promising candidate in breast cancer therapy due to its ability to modulate key oncogenic pathways. Its mechanisms of action include the inhibition of cyclooxygenase (COX) enzymes, which mitigates tumor-promoting inflammation and fosters a less permissive microenvironment for cancer progression. Additionally, talniflumate disrupts ionic homeostasis by targeting calcium-activated chloride channels (CaCCs), leading to impaired cellular proliferation and potential induction of apoptosis. The agent also exhibits anti-angiogenic activity by downregulating vascular endothelial growth factor (VEGF), thereby restricting tumor vascularization and growth. Furthermore, talniflumate shows potential as a chemosensitizer, enhancing the cytotoxic effects of standard chemotherapy and improving therapeutic outcomes while reducing chemoresistance. These multifaceted mechanisms highlight the therapeutic promise of talniflumate in breast cancer, warranting further preclinical and clinical studies to validate its efficacy, refine dosing strategies, and define its role in combination therapies.

PURPOSE:

To assess the therapeutic efficacy of Talniflumate in the management of breast cancer, with a focus on its synergistic interactions with neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 and ≤ 75 years, female;
* The breast cancer has been confirmed by pathological examination and Immunohistochemistry (IHC);
* Not receiving any preoperative anticancer drugs;
* The liver and kidney function satisfies the following conditions within 3 days after surgery (excluding day 3): aspartate aminotransferase (AST), glutamic-oxalacetic transaminase (ALT) < 2 upper limit of normal (ULN), total bilirubin ≤ 1.5 ULN, serum creatinine < 1.5 ULN;
* Other laboratory tests meet the following requirements within 3 days after surgery (excluding day 3): Hb ≥ 90g/l, platelet count ≥ 100×109/L, absolute neutrophil count > 1.5×109/L;
* The expected survival time ≥ 6 months;
* The subjects volunteer to sign the informed consent.

Exclusion Criteria:

* Patients with stage IV breast cancer;
* Pregnant or lactating women;
* Those with active bleeding due to various reasons;
* Those with HIV infection or AIDS-associated diseases;
* Those with severe acute and chronic diseases;
* Those with severe diabetes;
* Those with serious infectious diseases;
* Those who can not take drugs by oral route;
* Drug abusers or those with psychological or mental diseases that may interfere with study compliance;
* Conditions that are considered not suitable for this study investigators

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Up to 5 years
  Time from randomization to recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first, assessed up to 5 years.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Time from randomization to death from any cause, assessed up to 5 years.

REFERENCES:
- [Background] Wang X, Chen B, Zhang H, Peng L, Liu X, Zhang Q, Wang X, Peng S, Wang K, Liao L. Integrative analysis identifies molecular features of fibroblast and the significance of fibrosis on neoadjuvant chemotherapy response in breast cancer. Int J Surg. 2024 Jul 1;110(7):4083-4095. doi: 10.1097/JS9.0000000000001360. PMID 38546506
- [Background] Spanheimer PM, Reeder-Hayes KE. Breast surgery after neoadjuvant chemotherapy: time for a change? Lancet Oncol. 2022 Dec;23(12):1477-1479. doi: 10.1016/S1470-2045(22)00649-0. Epub 2022 Oct 25. No abstract available. PMID 36306811
- [Background] Rao CV, Janakiram NB, Madka V, Kumar G, Scott EJ, Pathuri G, Bryant T, Kutche H, Zhang Y, Biddick L, Gali H, Zhao YD, Lightfoot S, Mohammed A. Small-Molecule Inhibition of GCNT3 Disrupts Mucin Biosynthesis and Malignant Cellular Behaviors in Pancreatic Cancer. Cancer Res. 2016 Apr 1;76(7):1965-74. doi: 10.1158/0008-5472.CAN-15-2820. Epub 2016 Feb 15. PMID 26880801
- [Background] Agostini A, Guerriero I, Piro G, Quero G, Roberto L, Esposito A, Caggiano A, Priori L, Scaglione G, De Sanctis F, Sistigu A, Musella M, Larghi A, Rizzatti G, Lucchetti D, Alfieri S, Sgambato A, Bria E, Bizzozero L, Arena S, Ugel S, Corbo V, Tortora G, Carbone C. Talniflumate abrogates mucin immune suppressive barrier improving efficacy of gemcitabine and nab-paclitaxel treatment in pancreatic cancer. J Transl Med. 2023 Nov 23;21(1):843. doi: 10.1186/s12967-023-04733-z. PMID 37996891